CLINICAL TRIAL: NCT01208649
Title: Effects of Exenatide (Byetta®) on Biochemical and Histological Parameters of Liver Function in Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: Effects of Exenatide (Byetta®) on Liver Function in Patients With Nonalcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Prof. Dr. med. Wolfgang E. Schmidt; Director Department of Medicine l;, Universitiy Hospital; Ruhr-University Bochum; Gudrunstr. 56; 44791 Bochum; Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H80-MC-O008
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: exenatide; hepatic steatosis; insulin resistance; insulin sensitizers; nonalcoholic fatty liver disease; - GLP1-Analog
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver; Insulin Resistance | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Active Comparator): Drug (including placebo)
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide; 48 weeks 10 microg injection s.c., twice daily, before the morning and evening meal with a four week wash-in phase with 5 microg injection s.c.twice daily

SUMMARY:
The primary objective is to test the hypothesis that 24 weeks of treatment with exenatide will improve the histological acitvity of NASH (steatosis,necroinflammation, ballooning), summarized in the recently introduced NASH-score in patients with normal, impaired or diabetic glucose tolerance compared to dietary guidance alone.

DETAILED DESCRIPTION:
Non alcoholic steatohepatitis (NASH), a chronic liver disease characterized by insulin resistance, accumulation of hepatic fat and hepatocellular necroinflammation, has been recognized as a leading cause of (cryptogenic) liver cirrhosis in developed countries. Given the rising prevalence of NASH and the associated socio-economic burden associated, novel therapeutic options are warranted. The incretin mimetic Exenatide (Byetta®) exhibits strong glucoregulatory activities through its multiple biological effects. In addition, exenatide treatment has been shown to improve lipid homeostasis and reduce body weight. Since the development of NASH has been tightly linked to the presence of obesity, hyperlipidaemia and diabetes, this study will examine, whether 24 weeks of treatment with exenatide will also result in improvements in liver function in patients with NASH.

60 patients with histologically proven NASH will be randomized to receive either exenatide (2 x 5 µg s.c. for 4 weeks, 2 x 10 µg thereafter) or placebo treatment, in a 1:1 ratio. Liver biopsies will be performed after 24 weeks of treatment. In addition, a non-invasive assessment of hepatic mitochondrial function will be carried-out using a 13C-methionine breath test at baseline, and at weeks 12 and 24. Insulin sensitivity and glucose tolerance will be assessed by a hyperinsulinaemic-euglycaemic clamp (baseline and week 24) and an oral glucose tolerance test (baseline, weeks 12 and 24). Hepatic fat content will be measured by magnetic resonance tomography. Liver enzymes will be monitored closely throughout the study period.

These studies will clarify whether exenatide treatment, in addition to its beneficial effects on glucose homeostasis and body weight, will also result in improvements of liver function in patients with NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, inclusive.
2. Patients present with histologically proven non-alcoholic steatohepatitis ascertained by the single center pathologist between visit 1 and 2
3. First liver biopsy was obtained not later than 6 months before visit 1
4. Patients have HbA1c not exceeding 10.0%.
5. Patients have a history of stable body weight (not varying by >10% for at least 3 months prior to screening

Exclusion Criteria:

1. Patients are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
2. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomised partner). A male subject who is sexually active and has not been surgically sterilised must be informed that he must either use a condom during intercourse, ensure that his partner practices contraception, or he must refrain from sexual intercourse during the trial and until 1 month after completion of the trial. This is to prevent the possibility of a pregnancy from spermatocytes that can potentially be damaged by trial medication. It is strongly recommended that the female partners use a highly effective contraception (Pearl Index < 1%).
3. Patients have participated in an interventional medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment was given) within 30 days prior to screening. This criterion includes drugs that have not received regulatory approval for any indication at the time of study entry.
4. Patients with evidence of viral or autoimmune hepatitis (positive testing for HBsAG, anti-HCV or anti-HIV, pos. AMA-screen, ANA-titer > 1:160)
5. Patients with inherited liver diseases (e.g. Wilson's disease, Hemochromatosis)
6. Patients have alcohol consumption (>20 g daily for males and >10 g daily for females)
7. Patients have decompensated liver cirrhosis (Child-Pugh score >7)
8. Patients have alanine aminotransaminase (ALT) greater than ten times the upper limit of the reference range.
9. Patients have had greater than three episodes of severe hypoglycemia within 6 months prior to screening.
10. Patients are undergoing therapy for a malignancy, other than basal cell or squamous cell skin cancer.
11. Patients have cardiac disease that is Class III or IV, according to the New York Heart Association criteria.
12. Patients have a known allergy or hypersensitivity to exenatide, or excipients contained in these agents.
13. Patients have or had concomitant medication with thiazolidinediones.
14. Patients have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine >1.8 mg/dL for males and greater than or equal to >1.5 mg/dL for females.
15. Patients have known hemoglobinopathy or chronic anemia
16. Patients are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to screening.
17. Patients have used any prescription drug to promote weight loss within 3 months prior to screening.
18. Patients have any other condition (including known drug or alcohol abuse or psychiatric disorder) that precludes them from following and completing the protocol, in the opinion of the investigator.
19. Patients fail to satisfy the investigator of suitability to participate for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
histological activity of NASH (steatosis, necroinflammation, ballooning) | 24 weeks

SECONDARY OUTCOMES:
Liver fibrosis, as determined using the fibrosis score | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang E. Schmidt, Prof. Dr., Study Director — Ruhr-University Bochum; Wolfgang E. Schmidt, Prof. Dr., Principal Investigator — Ruhr-University Bochum
Locations (1):
- Department of Medicine I; University Hospital St. Josef-Hospital, Bochum, Germany